CLINICAL TRIAL: NCT06559826
Title: A Randomized-Controlled Trial of Ketamine-Assisted Psychotherapy (KAP) Compared to Ketamine Alone for the Treatment of Depression
Brief Title: Ketamine-Assisted Psychotherapy (KAP) Compared to Ketamine Alone for the Treatment of Depression
Acronym: KAP
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, James Murrough, Professor of Psychiatry and Neuroscience, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-23-00661; PD23-03701 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2024-08-15; First posted 2024-08-19 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder
Keywords: Ketamine; Major Depressive Disorder; Ketamine Assisted Psychotherapy
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Ketamine; Psychotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Assisted Psychotherapy (KAP) (Experimental): KAP sessions will occur once a week for a total of 4 weeks with the potential for a second session the first week for dose-finding purposes. Participants will have a ketamine exposure of at least 0.3 mg/kg and a maximum of 1.0mg/kg, at each treatment session, personalizing dose to patient experience. Each of the treatment sessions will last 120-180 min and will be conducted by a single therapist who has completed the KAP training as specified in the standard operating procedures.
  Interventions: Drug: Ketamine; Behavioral: Psychotherapy
- Ketamine (KET) (Active Comparator): Standard medicalized ketamine administration consisting of twice weekly treatment for 3 weeks, followed by a 4th week with a single ketamine infusion serving as a down-titration period before discontinuation. Participants will have a ketamine exposure of at least 0.3 mg/kg administered via intravenous infusion at each treatment session. Patients may be up-titrated over the course of subsequent treatment sessions, as indicated clinically up to 1.0 mg/kg25. No formal psychotherapy will be provided in the KET arm, though study participants will have matched basic psychoeducation related to depression and treatment with ketamine prior to the first dosing session, during the ketamine treatment period, and post-treatment, in order to match the KAP arm. All individuals will be followed over an eight week follow up period and undergo clinical study assessments.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Following screening and baseline assessments, individuals randomized to KAP will undergo a preparatory session prior to the first day of dosing. Participants will complete a sequence of four to five intramuscular (IM) ketamine assisted therapy sessions.
Behavioral: Psychotherapy — Each week following KAP, there will be a separate 60-minute integration session 1-6 days afterwards. Integration sessions will focus on processing experiences and material that emerged in KAP sessions (such as assimilating challenging experiences, making meaning of experiences and imagery, working through memories and emotions, and exploring emerging relational patterns) as well as strengthening insights. Within one week of the completion of all KAP sessions, there will be one additional integration session focused on consolidating the insights and improvements gained from KAP treatment.
  Arms: Ketamine Assisted Psychotherapy (KAP)

SUMMARY:
The proposed study is a single-site, randomized, controlled clinical trial (RCT) comparing ketamine-assisted psychotherapy (KAP) to a standard evidence-based regimen of ketamine administered in a medical model without psychotherapy (KET). Eligible study participants will be adults with major depressive disorder (MDD). Adults with MDD will be randomized to KAP or KET in a 1:1 allocation. Each treatment group will receive KAP or KET over a period of four weeks. Measurement of depression severity, wellness, neurocognitive functioning and other parameters will occur at baseline prior to treatment, immediately following the end of the acute treatment period, and over an 8-week (two month) treatment follow-up period.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent (and assent when applicable) obtained from subject and ability for subject to comply with the requirements of the study.
* Age 18-90 years
* Participant in good physical health
* Participants may be on medications for depression as long as they remain on a stable dose.
* A score of at least 20 on the 10 item Montgomery-Asberg Depression Scale at screening, corresponding to at least moderate current depression severity.
* Meets criteria for major depressive disorder (MDD) in current major depressive episode (MDE) according to DSM-5
* Women of child-bearing potential must have a negative pregnancy test at screening and prior to ketamine infusion

Exclusion Criteria

* Pregnant, breastfeeding, or unwilling to practice birth control during participation in the study.
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data.
* Any unstable medical illnesses including hepatic, renal, gastroenterological, respiratory, cardiovascular (including ischemic heart disease and uncontrolled hypertension); endocrinologic, neurologic, immunologic, or hematologic disease
* Clinically significant abnormalities of laboratories, physical examination, or ECG
* Substance drug or alcohol use disorder in the prior 12 months
* History of hypersensitivity to ketamine or esketamine
* Lifetime history of schizophrenia, schizoaffective disorder, bipolar I or II disorder
* Presence of psychotic symptoms in the current MDE, or lifetime psychotic disorder
* Recreational ketamine or phencyclidine use in the last year
* Previous non-response to clinical or research ketamine or esketamine administration
* Concurrent treatment with ECT, TMS, or VNS in the current MDE
* BMI > 35
* Significant suicidal ideation as determined by a C-SSRS score >2 in past 30 days
* History of suicide attempt or self harm in the prior 2 years
* SBP > 165 or DBP > 95 on infusion day
* MoCA score < 23

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | 9 weeks from baseline assessment
  MADRS: The Montgomery-Asberg Depression Rating Scale (MADRS) is a 10-item instrument used for the evaluation of depressive symptoms in adults and for the assessment of any changes to those symptoms. Each of the 10 items is rated on a scale of 0 to 6, with differing descriptors for each item. These individual item scores are added together to form a total score, which can range between 0 and 60 points, with higher scores indicating more severe depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: James Murrough, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
This is a study funded by private philanthropy and therefore we do not plan to share the results from the data.